Study Title: Feasibility of the Camp Power Up Program on Children's Body Weight and Quality of Life

NCT #: NCT03235440

Document date: September 1, 2020

We used SPSS to conduct paired t-tests to analyze any pre-to-posttest changes in health behaviors and psychosocial well-being outcomes. Cohen's d was computed as effect size to interpret the between time differences. Subsequently, we conducted repeated measure multivariate analyses of variance (RM-MANOVAs) to examine pre-to-posttest changes in health behaviors and psychosocial well-being outcomes by gender (boys vs. girls) and household income (\$50,000 as the split value). We further explored the pre-to-posttest changes in the outcomes (using gain scores: posttest — pretest data) by weight status (normal weight, overweight, obesity), but did not perform inferential statistical analysis due to the uneven sample sizes between the weight groups. Descriptive results including both raw and estimated marginal means were obtained to quantify and visualize group differences. Partial eta square () was reported as effect size from results from the RM-MANOVAs, while significance level was set to be  $\alpha = 0.05$ .